CLINICAL TRIAL: NCT05182268
Title: Comparison of Clinical Effect Between Endoscopic and Microscopic Ear Surgery of Cholesteatoma: A Multicenter Retrospective Observational Study
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SunYatsenU2H_YangH01
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Endoscopy; Microscopy; Ear Surgery; Cholesteatoma; Clinical Effect
MeSH Terms: conditions — Cholesteatoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- endoscopic ear surgery group(EES)
  Interventions: Procedure: endoscopic ear surgery
- microscopic ear surgery group(MES)
  Interventions: Procedure: microscopic ear surgery

INTERVENTIONS:
Procedure: endoscopic ear surgery — a ear surgery via endoscopic
  Groups: endoscopic ear surgery group(EES)
Procedure: microscopic ear surgery — a ear surgery via microscopic
  Groups: microscopic ear surgery group(MES)

SUMMARY:
Background: Cholesteatoma is a potentially life-threatening inflammatory lesion that causes hearing loss, ear discharge, and ear pain, and serious complications. For the past several decades, most studies of cholesteatoma have been restricted to microscopic ear surgery. However, a growing body of evidence suggests endoscopic ear surgery is a safe, minimally invasive approach for cholesteatoma management. This thesis aim to investigate and compare the clinical effect between endoscopic and microscopic ear surgery of cholesteatoma.

Materials and methods: The retrospective study included 186 patients with cholesteatoma who received endoscopic or microscopic ear surgery from 11 otorhinolaryngology centers between November 2016 and March 2021. Patients were followed-up for at least 1 year. Audiometry improvement, treatment cost, time, graft success rate and recurrence rate were assessed after surgery.

ELIGIBILITY:
Inclusion Criteria:

* postoperative pathologically were confirmed cholesteatoma with or without mastoid involvement
* the extent of disease was confirmed by preoperative HRCT temporal bone
* undergoed microscopic and/or endoscopic surgery for cholesteatoma including primary or revision surgery

Exclusion Criteria:

* were lacking in clinical characteristics
* had not preoperative audiometric data
* missed the follow-up data
* were lacking in surgical times
* were microscopic combined endoscopic ear surgery

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Patients who postoperative pathologically were confirmed cholesteatoma with or without mastoid involvement. The extent of disease was confirmed by preoperative HRCT temporal bone.
  2. The patients undergoed microscopic and/or endoscopic surgery for cholesteatoma including primary or revision surgery.
  3. have completely clinical characteristics, follow-up data and/or postoperative audiometric data
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Pure Tone Average(PTA) | at least 1 year
  estimate the auditory acuity
Air-Bone Gap(A-B Gap) | at least 1 year
  estimate the auditory acuity